CLINICAL TRIAL: NCT02014558
Title: A Phase 1/2 Open-Label, Dose Escalation Study Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ASP2215 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Dose Escalation Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of ASP2215 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0101
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2013-11-06; First posted 2013-12-18 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Gilteritinib; ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; Voriconazole; Midazolam; Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (13):
- Gilteritinib 20 mg in Escalation Phase (Experimental): Participants received a single dose of 20 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 20 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
  Interventions: Drug: Gilteritinib; Drug: Voriconazole
- Gilteritinib 40 mg in Escalation Phase (Experimental): Participants received a single dose of 40 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 40 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 80 mg in Escalation Phase (Experimental): Participants received a single dose of 80 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 80 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 120 mg in Escalation Phase (Experimental): Participants received a single dose of 120 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 120 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 200 mg in Escalation Phase (Experimental): Participants received a single dose of 200 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 200 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 300 mg in Escalation Phase (Experimental): Participants received a single dose of 300 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 300 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 450 mg in Escalation Phase (Experimental): Participants received a single dose of 450 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 450 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 20 mg in Expansion Phase (Experimental): Participants received 20 mg gilteritinib orally once daily stating on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. Starting on day 16 of cycle 1, participants also received 200 mg voriconazole orally every 12 hours through day 1 of cycle 2.
  Interventions: Drug: Gilteritinib
- Gilteritinib 40 mg in Expansion Phase (Experimental): Participants received 40 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 80 mg in Expansion Phase (Experimental): Participants received 80 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 120 mg in Expansion Phase (Experimental): Participants received 120 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
  Interventions: Drug: Gilteritinib
- Gilteritinib 200 mg in Expansion Phase (Experimental): Participants received 200 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. On day -1 and day 15 of cycle 1, certain participants also received 500 mg cephalexin as a single oral dose.
  Interventions: Drug: Gilteritinib; Drug: Cephalexin
- Gilteritinib 300 mg in Expansion Phase (Experimental): Participants received 300 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. On day -1 and day 15 of cycle 1, participants also received 2 mg midazolam as a single oral dose.
  Interventions: Drug: Gilteritinib; Drug: Midazolam

INTERVENTIONS:
Drug: Gilteritinib — Participants received gilteritinib oral tablets (10 mg, 40 mg or 100 mg, depending on the dose) once daily without food allowed for at least 2 hours before and 1 hour after dosing starting from day -2 and day of cycle 1, for continuous 28-day cycles.
  Other Names: ASP2215
Drug: Voriconazole — Participants received 200 mg voriconazole tablets daily every 12 hours starting from day 16 of cycle 1 through day 1 of cycle 2.
  Arms: Gilteritinib 20 mg in Escalation Phase
Drug: Midazolam — Participants received a single oral dose of 2 mg of midazolam syrup on day -1 and day 15 of cycle 1.
  Arms: Gilteritinib 300 mg in Expansion Phase
Drug: Cephalexin — Participants received a single oral dose of 500 mg cephalexin tablet or capsule on day -1 and day 15 of cycle 1.
  Arms: Gilteritinib 200 mg in Expansion Phase

SUMMARY:
The objective of this study was to assess the safety and tolerability, including the maximum tolerated dose, of gilteritinib in participants with relapsed or treatment-refractory acute myeloid leukemia (AML). This study also determined the pharmacokinetic (PK) parameters of gilteritinib.

ELIGIBILITY:
Inclusion Criteria:

* Subject is defined as morphologically documented primary or secondary AML by the World Health Organization (WHO) criteria (2008) and fulfills one of the following:

  * Refractory to at least 1 cycle of induction chemotherapy
  * Relapsed after achieving remission with a prior therapy
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Subject's interval from prior treatment to time of study drug administration is at least 2 weeks for cytotoxic agents (except hydroxyurea given for controlling blast cells), or at least 5 half-lives for prior experimental agents or noncytotoxic agents.
* Subject must meet the following criteria as indicated on the clinical laboratory tests*:

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x institutional upper limit normal (ULN)
  * Total serum bilirubin < 1.5x institutional ULN
  * Serum creatinine < 1.5 x institutional ULN or an estimated glomerular filtration rate (eGFR) of > 50 ml/min as calculated by the Modification of Diet in Renal Disease (MDRD) equation.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject was diagnosed as acute promyelocytic leukemia (APL).
* Subject has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has active malignant tumors other than AML or Myelodysplastic syndrome (MDS).
* Subject has persistent nonhematological toxicities of >= Grade 2 (Common Terminology Criteria for Adverse Events v4), with symptoms and objective findings, from prior AML treatment (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, radiation, or surgery).
* Subject has had hematopoietic stem cell transplant (HSCT) and meets any of the following:

  * Is within 2 months of transplant from C1D1
  * Has clinically significant graft-versus-host disease requiring treatment
  * Has >= Grade 2 persistent non-hematological toxicity related to the transplant. Donor lymphocytes infusion (DLI) is not permitted <= 30 days prior to study registration or during the first cycle of treatment on the study in Cohort 1 and first two cycles of the treatment in Cohort 2
* Subject has clinically active central nervous system leukemia
* Subject has disseminated intravascular coagulation abnormality (DIC)
* Subject has had major surgery within 4 weeks prior to the first study dose.
* Subject has had radiation therapy within 4 weeks prior to the first study dose
* Subject has congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subject with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 3 months prior to study entry results in a left ventricular ejection fraction that is ≥ 45%
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of Cytochrome P450-isozyme3A4 (CYP3A4) with the exception of antibiotics, antifungals, and antivirals that are used as standard of care post-transplant or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the subject
* Subject required treatment with concomitant drugs that target serotonin 5HT1R or 5HT2BR receptors or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject has an active uncontrolled infection
* Subject is known to have human immunodeficiency virus infection
* Subject has active hepatitis B or C, or other active hepatic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development
Locations (26):
- United States (23):
  - Site US10021, Birmingham, Alabama
  - Site US10023, Scottsdale, Arizona
  - Site US10022, Duarte, California
  - Site US10008, Los Angeles, California
  - Site US10005, San Francisco, California
  - Site US10001, Chicago, Illinois
  - Site US10015, Chicago, Illinois
  - Site US10012, Baltimore, Maryland
  - Site US10003, Baltimore, Maryland
  - Site US10006, Minneapolis, Minnesota
  - Site US10011, Rochester, Minnesota
  - Site US10020, Hackensack, New Jersey
  - Site US10010, Buffalo, New York
  - Site US10009, New York, New York
  - Site US10013, New York, New York
  - Site US10019, New York, New York
  - Site US10014, Cleveland, Ohio
  - Site US10018, Hershey, Pennsylvania
  - Site US10004, Philadelphia, Pennsylvania
  - Site US10017, Charleston, South Carolina
  - Site US10007, Nashville, Tennessee
  - Site US10002, Houston, Texas
  - Site US10026, Fairfax, Virginia
- Germany (2):
  - Site DE49002, Berlin
  - Site DE49004, Dresden
- Site IT39001, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] James AJ, Smith CC, Litzow M, Perl AE, Altman JK, Shepard D, Kadokura T, Souda K, Patton M, Lu Z, Liu C, Moy S, Levis MJ, Bahceci E. Pharmacokinetic Profile of Gilteritinib: A Novel FLT-3 Tyrosine Kinase Inhibitor. Clin Pharmacokinet. 2020 Oct;59(10):1273-1290. doi: 10.1007/s40262-020-00888-w. PMID 32304015
- [Derived] Perl AE, Altman JK, Cortes J, Smith C, Litzow M, Baer MR, Claxton D, Erba HP, Gill S, Goldberg S, Jurcic JG, Larson RA, Liu C, Ritchie E, Schiller G, Spira AI, Strickland SA, Tibes R, Ustun C, Wang ES, Stuart R, Rollig C, Neubauer A, Martinelli G, Bahceci E, Levis M. Selective inhibition of FLT3 by gilteritinib in relapsed or refractory acute myeloid leukaemia: a multicentre, first-in-human, open-label, phase 1-2 study. Lancet Oncol. 2017 Aug;18(8):1061-1075. doi: 10.1016/S1470-2045(17)30416-3. Epub 2017 Jun 20. PMID 28645776
- [Derived] Kasi PM, Litzow MR, Patnaik MM, Hashmi SK, Gangat N. Clonal evolution of AML on novel FMS-like tyrosine kinase-3 (FLT3) inhibitor therapy with evolving actionable targets. Leuk Res Rep. 2016 Jan 12;5:7-10. doi: 10.1016/j.lrr.2016.01.002. eCollection 2016. PMID 26904404
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This dose-escalation/dose-expansion study was conducted in sites in the United States, France, Germany and Italy. The study had 7 dose-escalation cohorts with ≥3 participants enrolled at each dose level. Following escalation to the next dose cohort, additional participants were enrolled to the dose-expansion cohorts per protocol-specified criteria.
Pre-assignment Details: Participants with acute myeloid leukemia (AML) who relapsed after or were refractory to induction or salvage treatment were selected for this study. Five participants were re-enrolled into the dose-expansion cohorts as they discontinued treatment for reasons other than toxicity or disease progression, as long as they met the eligibility criteria.
Period: Overall Study
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase | Gilteritinib 20 mg in Expansion Phase | Gilteritinib 40 mg in Expansion Phase | Gilteritinib 80 mg in Expansion Phase | Gilteritinib 120 mg in Expansion Phase | Gilteritinib 200 mg in Expansion Phase | Gilteritinib 300 mg in Expansion Phase
Started (Re-enrolled participants (assigned to the 120 mg [1] & 200 mg [4] expansion groups) were excluded.) | 5 | 3 | 3 | 3 | 4 | 3 | 4 | 11 | 15 | 21 | 69 | 102 | 17
Treated | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 12 (A participant randomized to the 120 mg was treated with an initial dose of 20 mg by mistake.) | 13 | 21 | 66 (A participant randomized to the 120 mg was treated with an initial dose of 20 mg by mistake.) | 100 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 3 | 3 | 3 | 4 | 3 | 4 | 11 | 15 | 21 | 69 | 102 | 17
Not completed — Never Received Study Drug | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 5 | 21 | 3
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 5 | 5 | 19 | 2
Not completed — Lack of Efficacy | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 3 | 3 | 3 | 16 | 8 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 6 | 5 | 6 | 22 | 31 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 6 | 10 | 0
Not completed — Miscellaneous | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 12 | 11 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was the safety analysis set (SAF), which consisted of all participants who received at least 1 dose of study drug and excluded re-enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase | Gilteritinib 20 mg in Expansion Phase | Gilteritinib 40 mg in Expansion Phase | Gilteritinib 80 mg in Expansion Phase | Gilteritinib 120 mg in Expansion Phase | Gilteritinib 200 mg in Expansion Phase | Gilteritinib 300 mg in Expansion Phase | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 13 | 21 | 66 | 100 | 17 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (6.8) | 56.7 (6.7) | 61 (8.7) | 61.7 (6) | 64 (1) | 55.3 (25) | 61.7 (10.7) | 59.3 (15.6) | 59.6 (14) | 56.3 (18.1) | 58.3 (16.7) | 59.8 (14.6) | 57.7 (15.9) | 59 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 8 | 4 | 12 | 37 | 49 | 5 | 123
  Male | 3 | 2 | 2 | 2 | 1 | 2 | 3 | 4 | 9 | 9 | 29 | 51 | 12 | 129
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4 | 2 | 4 | 3 | 16
  White | 5 | 2 | 3 | 2 | 1 | 3 | 3 | 10 | 9 | 14 | 57 | 91 | 13 | 213
  Asian | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 7
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 6 | 1 | 1 | 16
Ethnicity [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 5 | 3 | 2 | 3 | 3 | 3 | 3 | 11 | 12 | 20 | 62 | 97 | 17 | 241
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 3 | 0 | 11
Duration of Disease (AML) [Mean (Standard Deviation); unit: months] — Population: The analysis population was the SAF, with participants with data available.
  months
    number analyzed (Participants) | 4 | 3 | 2 | 3 | 2 | 1 | 3 | 10 | 11 | 17 | 46 | 77 | 15 | 194
    (all) | 19.70 (24.62) | 10.81 (8.58) | 62.46 (6.97) | 49.53 (72.17) | 9.46 (2.23) | 19.75 (NA) — Data could not be calculated as there is only one participant in this arm who had available data. | 7.21 (4.27) | 11.3 (6.61) | 10.53 (11.22) | 16.3 (9.85) | 12.65 (11.33) | 10.9 (9.94) | 12.09 (17.76) | 13.16 (14.97)
Local FLT3 Mutation Status [Count of Participants; unit: Participants]
  Negative | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 8 | 12 | 13 | 10 | 9 | 58
  Positive | 4 | 3 | 3 | 2 | 2 | 2 | 2 | 11 | 5 | 9 | 53 | 90 | 8 | 194

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: To determine the maximum tolerated dose, safety was assessed by DLTs, defined as any grade ≥ 3 non-hematologic or extramedullary toxicity that occurred within 30 days starting with the first dose taken on day -2, and included the first treatment cycle in the dose escalation phase and in the first treatment cycle (28 days) in the dose expansion phase, that was considered to be possibly or probably related to study drug. Exceptions to this were the following: (1) Alopecia, anorexia or fatigue, (2) Grade 3 nausea and/or vomiting if not required tube feeding or total parenteral nutrition, or diarrhea if not required or prolonged hospitalization that was managed to grade ≤ 2 with standard antiemetic or antidiarrheal medications used at prescribed dose within 7 days of onset, (3) Grade 3 fever with neutropenia, with or without infection, (4) Grade 3 infection.
Time Frame: From first dose up to end of cycle 1 (30 days)
Population: The analysis population was the SAF. Only evaluable participants (defined as participants who received at least 80% of the intended dose during cycle 1 [received at least 23 daily doses in escalation phase or 22 daily doses in expansion phase during cycle 1] or participants who developed DLT within cycle 1) were included.
Measure: Count of Participants; unit: Participants
Groups:
- Gilteritinib 120 mg in Escalation Phase: Participants received a single dose of 120 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 120 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
- Gilteritinib 40 mg in Expansion Phase: Participants received 40 mg gilteritinib orally once daily stating on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
- Gilteritinib 80 mg in Expansion Phase: Participants received 80 mg gilteritinib orally once daily stating on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
- Gilteritinib 120 mg in Expansion Phase: Participants received 120 mg gilteritinib orally once daily stating on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
- Gilteritinib 200 mg in Expansion Phase: Participants received 200 mg gilteritinib orally once daily stating on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. On day -1 and day 15 of cycle 1, certain participants also received 500 mg cephalexin as a single oral dose.
- Gilteritinib 300 mg in Expansion Phase: Participants received 300 mg gilteritinib orally once daily stating on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. On day -1 and day 15 of cycle 1, participants also received 2 mg midazolam as a single oral dose.
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase | Gilteritinib 20 mg in Expansion Phase | Gilteritinib 40 mg in Expansion Phase | Gilteritinib 80 mg in Expansion Phase | Gilteritinib 120 mg in Expansion Phase | Gilteritinib 200 mg in Expansion Phase | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 11 | 18 | 62 | 87 | 13
Participants
  Any DLT | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 7 | 15 | 3
  Blood and lymphatic system disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cardiac disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Eye disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Gastrointestinal disorders | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 1
  General disorders & administration site conditions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hepatobiliary disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections and infestations | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Investigations | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 6 | 2
  Metabolism and nutrition disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Musculoskeletal and connective tissue disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Nervous system disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
  Renal and urinary disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Reproductive system and breast disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
  Vascular disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety was assessed by AEs, which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A treatment-emergent AE (TEAE) was defined as an AE observed after starting administration of the study drug up to 30 days after last dose of study drug (for participants who underwent hematopoietic stem cell transplantation [HSCT]: defined as AEs observed after starting study drug until the last dose before on study HSCT plus 30 days, and AEs that began after resumption of gilteritinib and within 30 days after the last dose of gilteritinib). AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (1-Mild, 2-Moderate, 3-Severe, 4-LifeThreatening, 5-Death).
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase | Gilteritinib 20 mg in Expansion Phase | Gilteritinib 40 mg in Expansion Phase | Gilteritinib 80 mg in Expansion Phase | Gilteritinib 120 mg in Expansion Phase | Gilteritinib 200 mg in Expansion Phase | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 13 | 21 | 66 | 100 | 17
Participants
  AEs | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 13 | 20 | 64 | 100 | 17
  Drug-Related AEs | 3 | 2 | 1 | 3 | 3 | 2 | 3 | 7 | 6 | 17 | 52 | 77 | 13
  Deaths | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 3 | 4 | 11 | 23 | 49 | 7
  Serious AEs | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 8 | 12 | 19 | 52 | 92 | 14
  Drug-Related Serious AEs | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 10 | 19 | 36 | 4
  AEs Leading to Discontinuation of Study Drug | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 5 | 11 | 12 | 46 | 6
  Drug-Related AEs Leading to Discont. of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 5 | 10 | 3
  Grade 3 or Higher TEAEs | 3 | 2 | 2 | 1 | 2 | 2 | 3 | 9 | 13 | 20 | 59 | 99 | 14
  AEs During On-Study HSCT Period | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 0
  Serious AEs During On-Study HSCT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0

3. Primary Outcome: Area Under the Concentration-time Curve Over the 24-Hour Dosing Interval (AUC24) After Single and Multiple Doses of Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -2 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose
Population: Pharmacokinetics analysis set (PKAS) - consisted of the subset of the SAF for which sufficient plasma concentration data were available to facilitate derivation of at least 1 pharmacokinetic parameter and for whom the time of dosing on the day of sampling was known. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 3 | 3
ng*h/mL
  Day -2: number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 3 | 2
  Day -2 | 302.1 (207.0) | 360.0 (223.5) | 1216 (472.6) | 2480 (1972) | 3022 (843.6) | 4163 (3178) | 3324 (221.1)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3 | 1
  Cycle 1 Day 15 | 1299 (1006) | 2482 (33.28) | 6958 (3273) | 6943 (3221) | 31428 (21412) | 31005 (10068) | 34768 (NA) — This cannot be calculated due to insufficient data (only 1 participant had available data).
Statistical Analysis 1: Comparison: Gilteritinib 20 mg in Escalation Phase vs Gilteritinib 40 mg in Escalation Phase vs Gilteritinib 80 mg in Escalation Phase vs Gilteritinib 120 mg in Escalation Phase vs Gilteritinib 200 mg in Escalation Phase vs Gilteritinib 300 mg in Escalation Phase vs Gilteritinib 450 mg in Escalation Phase; Dose Proportionality (Single Dose / Day -2) was evaluated using the power model; Test type: Other; Slope = 0.990, 90% CI 2-sided [0.788 to 1.19]
Statistical Analysis 2: Comparison: Gilteritinib 20 mg in Escalation Phase vs Gilteritinib 40 mg in Escalation Phase vs Gilteritinib 80 mg in Escalation Phase vs Gilteritinib 120 mg in Escalation Phase vs Gilteritinib 200 mg in Escalation Phase vs Gilteritinib 300 mg in Escalation Phase vs Gilteritinib 450 mg in Escalation Phase; Dose Proportionality (Multiple Dose / Cycle 1 Day 15) was evaluated using the power model; Test type: Other; Slope = 1.22, 90% CI 2-sided [1.00 to 1.43]

4. Primary Outcome: Maximum Concentration (Cmax) After Single and Multiple Doses of Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -2 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose
Population: The analysis population was the PKAS with available data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 3 | 3
ng/mL
  Day -2 | 28.13 (21.49) | 24.98 (14.58) | 75.29 (25.22) | 136.7 (94.37) | 168.2 (45.34) | 204.3 (136.4) | 207.6 (51.81)
  Cycle 1 day 15: number analyzed (Participants) | 4 | 3 | 3 | 3 | 2 | 3 | 1
  Cycle 1 day 15 | 64.64 (48.77) | 107.6 (31.92) | 376.4 (150.5) | 374.2 (190.1) | 1462 (815.1) | 1525 (664.6) | 1528 (NA) — This cannot be calculated due to insufficient data (only 1 participant had available data).
Statistical Analysis 1: Comparison: Gilteritinib 20 mg in Escalation Phase vs Gilteritinib 40 mg in Escalation Phase vs Gilteritinib 80 mg in Escalation Phase vs Gilteritinib 120 mg in Escalation Phase vs Gilteritinib 200 mg in Escalation Phase vs Gilteritinib 300 mg in Escalation Phase vs Gilteritinib 450 mg in Escalation Phase; Dose Proportionality (Single Dose / Day -2) was evaluated using the power model; Test type: Other; Slope = 0.808, 90% CI 2-sided [0.629 to 0.988]
Statistical Analysis 2: Comparison: Gilteritinib 20 mg in Escalation Phase vs Gilteritinib 40 mg in Escalation Phase vs Gilteritinib 80 mg in Escalation Phase vs Gilteritinib 120 mg in Escalation Phase vs Gilteritinib 200 mg in Escalation Phase vs Gilteritinib 300 mg in Escalation Phase vs Gilteritinib 450 mg in Escalation Phase; Dose Proportionality (Multiple Dose / Cycle 1 Day 15) was evaluated using the power model; Test type: Other; Slope = 1.21, 90% CI 2-sided [1.02 to 1.41]

5. Primary Outcome: Area Under the Concentration-time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) After Single and Multiple Doses of Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -2 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose
Population: The analysis population was the PKAS with available data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 3 | 3
ng*h/mL
  Day -2 | 303.0 (207.1) | 360.4 (224.1) | 1216 (472.6) | 2480 (1972) | 3024 (846.2) | 4181 (3189) | 2544 (1427)
  Cycle 1 day -15: number analyzed (Participants) | 4 | 3 | 3 | 3 | 2 | 3 | 1
  Cycle 1 day -15 | 1030 (984.2) | 1990 (1422) | 7111 (3525) | 6943 (3221) | 32248 (22571) | 31749 (10090) | 35506 (NA) — This cannot be calculated due to insufficient data (only 1 participant had available data).

6. Primary Outcome: Time to Observed Cmax (Tmax) After Single and Multiple Doses of Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -2 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose
Population: The analysis population was the PKAS with available data.
Measure: Median (Full Range); unit: hours
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 3 | 3
hours
  Day -2 | 2.00 [0.500 to 4.03] | 5.983 [3.97 to 24.0] | 4.000 [4.00 to 4.08] | 2.083 [2.00 to 3.83] | 5.233 [4.00 to 5.97] | 6.067 [4.08 to 24.1] | 5.783 [4.08 to 5.92]
  Cycle 1 day 15: number analyzed (Participants) | 4 | 3 | 3 | 3 | 2 | 3 | 1
  Cycle 1 day 15 | 4.008 [4.00 to 6.00] | 3.867 [0.50 to 6.00] | 4.333 [4.00 to 4.42] | 2.167 [1.95 to 5.75] | 6.033 [6.00 to 6.07] | 6.050 [4.08 to 6.07] | 5.933 [NA to NA] — This cannot be calculated due to insufficient data (only 1 participant had available data).

7. Primary Outcome: Terminal Elimination Half-life (t1/2) After Multiple Doses of Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose
Population: The analysis population was the PKAS with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3 | 0
hours | 62.14 (17.88) | 151.8 (129.2) | 86.11 (24.08) | 45.85 (18.83) | 141.9 (61.51) | 142.2 (55.04) |

8. Primary Outcome: Accumulation Ratio After Multiple Doses of Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose
Population: The analysis population was the PKAS with available data.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Gilteritinib 450 mg in Escalation Phase: Participants received a single dose of 450 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 450 mg gilteritinib orally once daily in in the escalation phase of the study.28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
Arm/Group | Gilteritinib 20 mg in Escalation Phase | Gilteritinib 40 mg in Escalation Phase | Gilteritinib 80 mg in Escalation Phase | Gilteritinib 120 mg in Escalation Phase | Gilteritinib 200 mg in Escalation Phase | Gilteritinib 300 mg in Escalation Phase | Gilteritinib 450 mg in Escalation Phase
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3 | 0
ratio | 4.259 (1.069) | 9.640 (7.754) | 5.693 (1.442) | 3.290 (1.118) | 9.041 (3.693) | 9.057 (3.303) |

9. Secondary Outcome: Percentage of Participants With Complete Remission (CR) During the First 2 Cycles
Description: CR was defined according to modified Cheson criteria (2003), using centrally evaluated myeloblast counts from bone marrow aspirate/biopsy assessments and centrally evaluated hematology results; if neither central bone marrow aspirate nor biopsy was available, myeloblast was imputed with locally evaluated bone marrow aspirate/biopsy assessments (derived response). Participants were classified as being in CR when they had bone marrow regenerating normal hematopoietic cells, achieved a morphologic leukemia-free state, had an absolute neutrophil count (ANC) > 1 x 10^9/L, platelet count ≥ 100 x 10^9/L, normal marrow differential with < 5% blasts, had been red blood cell (RBC) and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion), had no presence of Auer rods and no evidence of extramedullary leukemia, and blast counts in peripheral blood had been ≤ 2%. Exact 95% confidence interval was estimated using binomial distribution.
Time Frame: During the first 2 cycles (56 days)
Population: Full analysis set (FAS) - consisted of all participants who were enrolled, took at least 1 dose of study drug and who had at least 1 posttreatment data point. Re-enrolled participants and participants from one site due to concerns with this site's GCP compliance were excluded. Participants were summarized under planned reporting groups in the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Gilteritinib 20 mg: Participants received 20 mg gilteritinib orally once on day -2, and starting on day 1 of cycle 1, participants received 20 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
- Gilteritinib 40 mg: Participants received 40 mg gilteritinib orally once on day -2, and starting on day 1 of cycle 1, participants received 40 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
- Gilteritinib 80 mg: Participants received 80 mg gilteritinib orally once on day -2, and starting on day 1 of cycle 1, participants received 80 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
- Gilteritinib 120 mg: Participants received 120 mg gilteritinib orally once on day -2, and starting on day 1 of cycle 1, participants received 120 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
- Gilteritinib 200 mg: Participants received 200 mg gilteritinib orally once on day -2, and starting on day 1 of cycle 1, participants received 200 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
- Gilteritinib 300 mg: Participants received 300 mg gilteritinib orally once on day -2, and starting on day 1 of cycle 1, participants received 300 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
- Gilteritinib 450 mg: Participants received 450 mg gilteritinib orally once on day -2, and starting on day 1 of cycle 1, participants received 450 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation.
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 8.3 [0.2 to 38.5] | 3.6 [0.4 to 12.3] | 3.4 [0.7 to 9.5] | 10 [0.3 to 44.5] | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 50.0 [1.3 to 98.7] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 6.3 [0.2 to 30.2] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 4.2 [0.1 to 21.1] | 2.9 [0.3 to 9.9] | 3.0 [0.6 to 8.5] | 5.0 [0.1 to 24.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events.

10. Secondary Outcome: Percentage of Participants With CR During Treatment
Description: as for outcome 9
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 16.7 [2.1 to 48.4] | 12.5 [5.2 to 24.1] | 11.2 [5.5 to 19.7] | 10.0 [0.3 to 44.5] | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 50.0 [1.3 to 98.7] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 6.3 [0.2 to 30.2] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 8.3 [1.0 to 27.0] | 10.0 [4.1 to 19.5] | 10.0 [4.9 to 17.6] | 5.0 [0.1 to 54.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events.

11. Secondary Outcome: Percentage of Participants With CR With Incomplete Platelet Recovery (CRp)
Description: CRp was defined according to modified Cheson criteria (2003), using centrally evaluated myeloblast counts from bone marrow aspirate/biopsy assessments and centrally evaluated hematology results; if neither central bone marrow aspirate nor biopsy was available, myeloblast was imputed with locally evaluated bone marrow aspirate/biopsy assessments (derived response). Participants were classified as being in CRp when they achieved CR except for incomplete platelet recovery (< 100 x 10^9/L). Exact 95% confidence interval was estimated using the binomial distribution.
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 3.6 [0.4 to 12.3] | 9.0 [4.0 to 16.9] | 10.0 [0.3 to 44.5] | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 2.9 [0.3 to 9.9] | 8.0 [3.5 to 15.2] | 5.0 [0.1 to 24.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events.

12. Secondary Outcome: Percentage of Participants With CR With Incomplete Hematological Recovery (CRi)
Description: CRi was defined according to modified Cheson criteria (2003), using centrally evaluated myeloblast counts from bone marrow aspirate/biopsy assessments and centrally evaluated hematology results; if neither central bone marrow aspirate nor biopsy was available, myeloblast was imputed with locally evaluated bone marrow aspirate/biopsy assessments (derived response). Participants were classified as being in CRi when they fulfilled all the criteria for CR except for incomplete hematological recovery with residual neutropenia < 1 x 10^9/L with or without complete platelet recovery. RBC and platelet transfusion independence were not required. Exact 95% confidence interval was estimated using the binomial distribution.
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 7.1 [0.2 to 33.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 25.0 [5.5 to 57.2] | 30.4 [18.8 to 44.1] | 20.2 [12.4 to 30.1] | 10.0 [0.3 to 44.5] | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 16.7 [2.1 to 48.4] | 7.1 [0.2 to 33.9] | 9.1 [0.2 to 41.3] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 6.3 [0.2 to 30.2] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 20.8 [7.1 to 42.2] | 25.7 [16.0 to 37.6] | 19.0 [11.8 to 28.1] | 5.0 [0.1 to 24.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events.

13. Secondary Outcome: Percentage of Participants With Complete Remission With Partial Hematologic Recovery (CRh)
Description: CRh was defined according to modified Cheson criteria (2003), using centrally evaluated myeloblast counts from bone marrow aspirate/biopsy assessments and centrally evaluated hematology results; if neither central bone marrow aspirate nor biopsy was available, myeloblast was imputed with locally evaluated bone marrow aspirate/biopsy assessments (derived response). Participants were classified as being in CRh when they could not be classified as being in CR and had bone marrow blasts < 5% and partial hematologic recovery ANC >= 0.5 x 10^9/L and platelets >= 50 x 10^9/L. There should not be evidence of extramedullary leukemia. Exact 95% confidence interval was estimated using the binomial distribution. CRh was calculated only for participants who were FLT3 mutation positive.
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS, with participants who were FLT3 mutation positive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
percentage of participants | 7.1 [0.2 to 33.9] | 0 [0 to 0] | 8.3 [0.2 to 38.5] | 10.7 [4.0 to 21.9] | 7.9 [3.2 to 15.5] | 20.0 [2.5 to 55.6] | 0 [0 to 0]

14. Secondary Outcome: Percentage of Participants With Composite CR (CRc)
Description: CRc was defined according to modified Cheson criteria (2003), using centrally evaluated myeloblast counts from bone marrow aspirate/biopsy assessments and centrally evaluated hematology results; if neither central bone marrow aspirate nor biopsy was available, myeloblast was imputed with locally evaluated bone marrow aspirate/biopsy assessments (derived response). Participants were classified as being in CRc when they had achieved either CR, complete remission with incomplete platelet recovery (CRp, defined as had achieved CR except for incomplete platelet recovery (< 100 x 10^9/L) or complete remission with incomplete hematologic recovery (CRi, defined as had fulfilled all the criteria for CR except for incomplete hematological recovery with residual neutropenia < 1 x 10^9/L with or without complete platelet recovery; RBC platelet transfusion independence not required). Exact 95% confidence interval was estimated using the binomial distribution.
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 7.1 [0.2 to 33.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 41.7 [15.2 to 72.3] | 46.4 [33.0 to 60.3] | 40.4 [30.2 to 51.4] | 30.0 [6.7 to 65.2] | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 50.0 [1.3 to 98.7] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 16.7 [2.1 to 48.4] | 7.1 [0.2 to 33.9] | 9.1 [0.2 to 41.3] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 12.5 [1.6 to 38.3] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 29.2 [12.6 to 51.1] | 38.6 [27.2 to 51.0] | 37.0 [27.6 to 47.2] | 15.0 [3.2 to 37.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events.

15. Secondary Outcome: Percentage of Participants With Partial Remission (PR)
Description: PR was defined according to modified Cheson criteria (2003), using centrally evaluated myeloblast counts from bone marrow aspirate/biopsy assessments and centrally evaluated hematology results; if neither central bone marrow aspirate nor biopsy was available, myeloblast was imputed with locally evaluated bone marrow aspirate/biopsy assessments (derived response). Participants were classified as being in PR when they had bone marrow regenerating normal hematopoietic cells with evidence of peripheral recovery with no (or only a few regenerating) circulating blasts and with a decrease of at least 50% in the percentage of blasts in the bone marrow aspirate with the total marrow blasts between 5% and 25%. A value of less or equal than 5% blasts was also considered a PR if Auer rods were present. There should be no evidence of extramedullary leukemia. Exact 95% confidence interval was estimated using the binomial distribution.
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 7.1 [0.2 to 33.9] | 37.5 [8.5 to 75.5] | 25.0 [5.5 to 57.2] | 7.1 [2.0 to 17.3] | 7.9 [3.2 to 15.5] | 30.0 [6.7 to 65.2] | 50.0 [1.3 to 98.7]
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 7.1 [0.2 to 33.9] | 9.1 [0.2 to 41.3] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 6.3 [0.2 to 30.2] | 18.8 [4.0 to 45.6] | 12.5 [2.7 to 32.4] | 7.1 [2.4 to 15.9] | 8.0 [3.5 to 15.2] | 15.0 [3.2 to 37.9] | 33.3 [0.8 to 90.6]

16. Secondary Outcome: Percentage of Participants With Best Response
Description: Best response was defined according to modified Cheson criteria (2003), using centrally evaluated myeloblast counts from bone marrow aspirate/biopsy assessments and centrally evaluated hematology results; if neither central bone marrow aspirate nor biopsy was available, myeloblast was imputed with locally evaluated bone marrow aspirate/biopsy assessments (derived response). BR was defined as the best measured response for all visits (in the order of CR, CRp, CRi, and PR) post-treatment. Participants who achieved the best response of CR, CRp, CRi or PR were classified as responders. Participants who did not achieve at least PR were considered as non-responders. Exact 95% confidence interval was estimated using the binomial distribution.
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 14.3 [1.8 to 42.8] | 37.5 [8.5 to 75.5] | 66.7 [34.9 to 90.1] | 53.6 [39.7 to 67.0] | 48.3 [37.6 to 59.2] | 60.0 [26.2 to 87.8] | 50.0 [1.3 to 98.7]
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 50.0 [1.3 to 98.7] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 16.7 [2.1 to 48.4] | 14.3 [1.8 to 42.8] | 18.2 [2.3 to 51.8] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 18.8 [4.0 to 45.6] | 18.8 [4.0 to 45.6] | 41.7 [22.1 to 63.4] | 45.7 [33.7 to 58.1] | 45.0 [35.0 to 55.3] | 30.0 [11.9 to 54.3] | 33.3 [0.8 to 90.6]

17. Secondary Outcome: Percentage of Participants With Complete Remission and Complete Remission With Partial Hematologic Recovery (CR/CRh)
Description: Participants with CR/CRh were defined as participants who achieved either CR or CRh. Participants with CR had bone marrow regenerating normal hematopoietic cells, achieved a morphologic leukemia-free state, had an ANC > 1 x 10^9/L, platelet count ≥ 100 x 10^9/L, and normal marrow differential with < 5% blasts, had been RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). Also, there had been no presence of Auer rods, no evidence of extramedullary leukemia, and blast counts in peripheral blood had been ≤ 2%. Participants with CRh could not be classified as being in CR and had bone marrow blasts < 5%, partial hematologic recovery ANC >= 0.5 x 10^9/L and platelets >= 50 x 10^9/L. There should not be evidence of extramedullary leukemia. Exact 95% confidence interval was estimated using the binomial distribution. CR/CRh was calculated only for participants who were FLT3 mutation positive.
Time Frame: Up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS, with participants who were FLT3 mutation positive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
percentage of participants | 7.1 [0.2 to 33.9] | 0 [NA to NA] — Data could not be calculated due to the low number of events. | 25.0 [5.5 to 57.2] | 23.2 [13.0 to 36.4] | 19.1 [11.5 to 28.8] | 30.0 [6.7 to 65.2] | 0 [NA to NA] — Data could not be calculated due to the low number of events.

18. Secondary Outcome: Duration of CR (DCR)
Description: DCR was defined as the time from the date of first CR until the date of documented relapse for participants who achieved CR. Participants who died without report of relapse were considered non-events and censored at their last relapse-free disease assessment date. Other participants who did not relapse on study were considered non-events and censored at the last relapse-free disease assessment date. DCR was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: From date of remission until end of study (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS. Only participants who achieved CR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 2 | 7 | 10 | 1 | 0
days
  FLT3 Mutation Positive: number analyzed (Participants) | 0 | 0 | 2 | 7 | 10 | 1 | 0
  FLT3 Mutation Positive |  |  | NA [NA to NA] — Data could not be calculated due to the low number of events. | NA [86.0 to NA] — Data could not be calculated due to the low number of events. | 419.0 [64.0 to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. |
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  FLT3 Mutation Negative | NA [NA to NA] — Data could not be calculated due to the low number of events. |  |  |  |  |  |
  All Participants | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | NA [NA to NA] — Data could not be calculated due to the low number of events. | NA [86.0 to NA] — Data could not be calculated due to the low number of events. | 419.0 [64.0 to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. |

19. Secondary Outcome: Duration of CRp (DCRp)
Description: DCRp was defined as the time from the date of first CRp until the date of documented relapse for participants who achieved CRp. Participants who died without report of relapse were considered non-events and censored at their last relapse-free disease assessment date. Other participants who did not relapse on study were considered non-events and censored at the last relapse-free disease assessment date. DCRp was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: as for outcome 18
Population: The analysis population was the FAS. Only participants who achieved CRp were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 0 | 0 | 1 | 6 | 12 | 2 | 0
days
  FLT3 Mutation Positive |  |  | NA [NA to NA] — Data could not be calculated due to the low number of events. | NA [57.0 to NA] — Data could not be calculated due to the low number of events. | 450.0 [43.0 to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. |
  FLT3 Mutation Negative: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  All Participants |  |  | NA [NA to NA] — Data could not be calculated due to the low number of events. | NA [57.0 to NA] — Data could not be calculated due to the low number of events. | 450.0 [43.0 to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. |

20. Secondary Outcome: Duration of CRi (DCRi)
Description: DCRi was defined as the time from the date of first CRi until the date of documented relapse for participants who achieved CRi. Participants who died without report of relapse and participants who did not relapse were considered non-events and censored at the last relapse-free disease assessment date. DCRi was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: as for outcome 18
Population: The analysis population was the FAS. Only participants who achieved CRi were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 7 | 24 | 31 | 1 | 0
days
  FLT3 Mutation Positive: number analyzed (Participants) | 1 | 0 | 5 | 23 | 30 | 1 | 0
  FLT3 Mutation Positive | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | NA [79.0 to NA] — Data could not be calculated due to the low number of events. | 120.0 [56.0 to 383.0] | 191.0 [57.0 to 420.0] | NA [NA to NA] — Data could not be calculated due to the low number of events. |
  FLT3 Mutation Negative: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0 | 0 | 0
  FLT3 Mutation Negative |  |  | 41.0 [22.0 to 60.0] | 99.0 [NA to NA] — Data could not be calculated due to the low number of events. |  |  |
  All Participants | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | 79.0 [22.0 to NA] — Data could not be calculated due to the low number of events. | 120.0 [58.0 to 383.0] | 191.0 [57.0 to 420.0] | NA [NA to NA] — Data could not be calculated due to the low number of events. |

21. Secondary Outcome: Duration of CRh (DCRh)
Description: DCRh was defined as the time from the date of first CRh until the date of documented relapse for participants who achieved CRh but did not have a best response of CR. Participants who died without report of relapse and participants who did not relapse were considered non-events and censored at the last relapse-free disease assessment date. DCRh was calculated using Kaplan-Meier method and therefore data are estimated. DCRh was calculated only for participants who were FLT3 mutation positive.
Time Frame: as for outcome 18
Population: The analysis population was the FAS. Only participants who achieved CRh were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 1 | 6 | 7 | 2 | 0
days | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | NA [NA to NA] — Data could not be calculated due to the low number of events. | 64.0 [18.0 to 85.0] | 101.0 [29.0 to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. |

22. Secondary Outcome: Duration of CRc (DCRc)
Description: DCRc was defined as the time from the date of first CRc until the date of documented relapse for participants who achieved CRc. Participants who died without report of relapse and participants who did not relapse were considered non-events and censored at the last relapse-free disease assessment date. DCRc was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: as for outcome 18
Population: The analysis population was the FAS. Only participants who achieved CRc were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 2 | 0 | 7 | 27 | 37 | 3 | 0
days
  FLT3 Mutation Positive: number analyzed (Participants) | 1 | 0 | 5 | 26 | 36 | 3 | 0
  FLT3 Mutation Positive | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | NA [79.0 to NA] — Data could not be calculated due to the low number of events. | 98.0 [57.0 to 307.0] | 191.0 [101.0 to 465.0] | NA [NA to NA] — Data could not be calculated due to the low number of events. |
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 2 | 1 | 1 | 0 | 0
  FLT3 Mutation Negative | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | 41.0 [22.0 to 60.0] | 99.0 [NA to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. |  |
  All Participants | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | 79.0 [22.0 to NA] — Data could not be calculated due to the low number of events. | 99.0 [58.0 to 307.0] | 191.0 [101.0 to 465.0] | NA [NA to NA] — Data could not be calculated due to the low number of events. |

23. Secondary Outcome: Duration of CR/CRh (DCRCRh)
Description: DCRCRh was defined as the time from the date of first DCRCRh until the date of documented relapse for participants who achieved CR or CRh. For participants who achieved both CR and CRh, the first CR date or CRh date, whichever occurred first, was used. Participants who died without report of relapse and participants who did not relapse were considered non-events and censored at the last relapse-free disease assessment date. DCRCRh was calculated using Kaplan-Meier method and therefore data are estimated. DCRCRh was calculated only for participants who were FLT3 mutation positive.
Time Frame: as for outcome 18
Population: The analysis population was the FAS. Only participants who achieved CR or CRh were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 3 | 13 | 17 | 3 | 0
days | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | NA [NA to NA] — Data could not be calculated due to the low number of events. | 307.0 [56.0 to NA] — Data could not be calculated due to the low number of events. | 308.0 [101.0 to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. |

24. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the date of either first CRc or PR until the date of documented relapse of any type for participants who achieved CRc or PR. Participants who died without report of relapse were considered non-events and censored at their last relapse-free disease assessment date. Other participants who did not relapse on study are considered non-events and censored at the last relapse-free assessment date. Duration of response was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: as for outcome 18
Population: The analysis population was the FAS. Only participants who achieved CRc or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 3 | 3 | 10 | 32 | 45 | 6 | 1
days
  FLT3 Mutation Positive: number analyzed (Participants) | 2 | 3 | 8 | 30 | 43 | 6 | 1
  FLT3 Mutation Positive | NA [NA to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. | 88.0 [9.0 to NA] — Data could not be calculated due to the low number of events. | 141.0 [58.0 to 383.0] | 220.0 [111.0 to 482.0] | 59.0 [15.0 to 59.0] | NA [NA to NA] — Data could not be calculated due to the low number of events.
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 2 | 2 | 2 | 0 | 0
  FLT3 Mutation Negative | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | 41.0 [22.0 to 60.0] | 109.5 [99.0 to 120.0] | 85.0 [NA to NA] — Data could not be calculated due to the low number of events. |  |
  All Participants | NA [NA to NA] — Data could not be calculated due to the low number of events. | NA [NA to NA] — Data could not be calculated due to the low number of events. | 79.0 [9.0 to NA] — Data could not be calculated due to the low number of events. | 126.0 [58.0 to 307.0] | 220.0 [85.0 to 482.0] | 59.0 [15.0 to 59.0] | NA [NA to NA] — Data could not be calculated due to the low number of events.

25. Secondary Outcome: Time to CR (TTCR)
Description: TTCR was defined as the time from the first dose of study drug until the date of first CR.
Time Frame: From first dose of study drug up to end of treatment (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Population: The analysis population was the FAS. Only participants who achieved CR were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 2 | 7 | 10 | 1 | 0
days
  FLT3 Mutation Positive: number analyzed (Participants) | 0 | 0 | 2 | 7 | 10 | 1 | 0
  FLT3 Mutation Positive |  |  | 171.5 [28 to 315] | 141.0 [29 to 364] | 93.0 [27 to 225] | 56.0 [56 to 56] |
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  FLT3 Mutation Negative | 30.0 [30 to 30] |  |  |  |  |  |
  All Participants | 30.0 [30 to 30] |  | 171.5 [28 to 315] | 141.0 [29 to 364] | 93.0 [27 to 225] | 56.0 [56 to 56] |

26. Secondary Outcome: Time to CRp (TTCRp)
Description: TTCRp was defined as the time from the first dose of study drug until the date of first CRp. TTCRp was evaluated for participants who achieved CRp.
Time Frame: as for outcome 25
Population: The analysis population was the FAS. Only participants who achieved CRp were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 0 | 0 | 1 | 6 | 12 | 2 | 0
days
  FLT3 Mutation Positive |  |  | 140.0 [140 to 140] | 195.0 [30 to 418] | 84.5 [28 to 392] | 29.0 [28 to 30] |
  FLT3 Mutation Negative: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  All Participants |  |  | 140.0 [140 to 140] | 195.0 [30 to 418] | 84.5 [28 to 392] | 29.0 [28 to 30] |

27. Secondary Outcome: Time to CRi (TTCRi)
Description: TTCRi was defined as the time from the first dose of study drug until the date of first CRi. TTCRi was evaluated for participants who achieved CRi.
Time Frame: as for outcome 25
Population: The analysis population was the FAS. Only participants who achieved CRi were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 7 | 24 | 31 | 1 | 0
days
  FLT3 Mutation Positive: number analyzed (Participants) | 1 | 0 | 5 | 23 | 30 | 1 | 0
  FLT3 Mutation Positive | 57.0 [57 to 57] |  | 57.0 [31 to 70] | 57.0 [26 to 170] | 39.5 [26 to 133] | 28.0 [28 to 28] |
  FLT3 Mutation Negative: number analyzed (Participants) | 0 | 0 | 2 | 1 | 1 | 0 | 0
  FLT3 Mutation Negative |  |  | 71.5 [71 to 72] | 30.0 [30 to 30] | 30.0 [30 to 30] |  |
  All Participants | 57.0 [57 to 57] |  | 64.0 [31 to 72] | 43.5 [26 to 170] | 35.0 [26 to 133] | 28.0 [28 to 28] |

28. Secondary Outcome: Time to First CR/CRh (TTFCRCRh)
Description: TTFCRCRh was defined as the time from the first dose of study drug until the date of first either CR or CRh. TTFCRCRh was evaluated for participants who achieved CR or CRh. For participants who achieve both CR and CRh, the first CR date or CRh date, whichever occurs first was used. TTFCRCRh was calculated only for participants who were FLT3 mutation positive.
Time Frame: as for outcome 25
Population: The analysis population was the FAS. Only participants who achieved CR or CRh were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 3 | 13 | 17 | 3 | 0
days | 57.0 [57 to 57] |  | 57.0 [28 to 140] | 59.0 [29 to 280] | 57.0 [27 to 245] | 28.0 [28 to 30] |

29. Secondary Outcome: Time to Best CR/CRh (TTBCRCRh)
Description: TTBCRCRh was defined as the time from the first dose of study drug until the first date that the best response of CR or CRh was achieved. TTBCRCRh was evaluated for participants who achieved CR or CRh. For participants who achieve both CR and CRh, the first CR date was used. TTBCRCRh was calculated only for participants who were FLT3 mutation positive.
Time Frame: as for outcome 25
Population: The analysis population was the FAS. Participants who achieved CR or CRh were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 1 | 0 | 3 | 13 | 17 | 3 | 0
days | 57.0 [57 to 57] |  | 57.0 [28 to 315] | 63.0 [29 to 364] | 88.0 [27 to 245] | 30.0 [28 to 56] |

30. Secondary Outcome: Time to CRc (TTCRc)
Description: TTCRc was defined as the time from the first dose of study drug until the date of first CRc. TTCRc was evaluated for participants who achieved CRc.
Time Frame: as for outcome 25
Population: The analysis population was the FAS. Only participants who achieved CRc were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 2 | 0 | 7 | 27 | 37 | 3 | 0
days
  FLT3 Mutation Positive: number analyzed (Participants) | 1 | 0 | 5 | 26 | 36 | 3 | 0
  FLT3 Mutation Positive | 57.0 [57 to 57] |  | 56.0 [28 to 64] | 30.0 [26 to 211] | 31.5 [26 to 197] | 28.0 [28 to 30] |
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 2 | 1 | 1 | 0 | 0
  FLT3 Mutation Negative | 30.0 [30 to 30] |  | 71.5 [71 to 72] | 30.0 [30 to 30] | 30.0 [30 to 30] |  |
  All Participants | 43.5 [30 to 57] |  | 57.0 [28 to 72] | 30.0 [26 to 211] | 31.0 [26 to 197] | 28.0 [28 to 30] |

31. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from the first dose of study drug until the date of either first CRc or PR. TTR was evaluated for participants who achieved CRc or PR.
Time Frame: as for outcome 25
Population: The analysis population was the FAS. Only participants who achieved CRc or PR were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 3 | 3 | 10 | 32 | 45 | 6 | 1
days
  FLT3 Mutation Positive: number analyzed (Participants) | 2 | 3 | 8 | 30 | 43 | 6 | 1
  FLT3 Mutation Positive | 61.5 [29 to 94] | 57.0 [31 to 64] | 31.0 [28 to 59] | 29.0 [26 to 211] | 29.0 [26 to 197] | 28.0 [26 to 61] | 31.0 [31 to 31]
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 2 | 2 | 2 | 0 | 0
  FLT3 Mutation Negative | 30.0 [30 to 30] |  | 71.5 [71 to 72] | 29.5 [29 to 30] | 29.5 [29 to 30] |  |
  All Participants | 30.0 [29 to 94] | 57.0 [31 to 64] | 43.5 [28 to 72] | 29.0 [26 to 211] | 29.0 [26 to 197] | 28.0 [26 to 61] | 31.0 [31 to 31]

32. Secondary Outcome: Time to Best Response (TTBR)
Description: TTBR was defined as the time from the first dose of study drug until the first disease assessment date when participant achieved best response. TTBR was evaluated in participants who achieved best response of CR, CRp, CRi, or PR.
Time Frame: as for outcome 25
Population: The analysis population was the FAS. Only participants who achieved CR, CRp, CRi, or PR were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 3 | 3 | 10 | 32 | 45 | 6 | 1
days
  FLT3 Mutation Positive: number analyzed (Participants) | 2 | 3 | 8 | 30 | 43 | 6 | 1
  FLT3 Mutation Positive | 75.5 [57 to 94] | 57.0 [31 to 64] | 44.0 [28 to 315] | 43.5 [26 to 364] | 57.0 [26 to 245] | 29.0 [26 to 61] | 31.0 [31 to 31]
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 2 | 2 | 2 | 0 | 0
  FLT3 Mutation Negative | 30.0 [30 to 30] |  | 71.5 [71 to 72] | 29.5 [29 to 30] | 29.5 [29 to 30] |  |
  All Participants | 57.0 [30 to 94] | 57.0 [31 to 64] | 58.0 [28 to 315] | 30.0 [26 to 364] | 56.0 [26 to 245] | 29.0 [26 to 61] | 31.0 [31 to 31]

33. Secondary Outcome: Overall Survival (OS)
Description: The time from the date of first dose of study drug until the date of death from any cause. For a participant who was not known to have died by the end of study follow-up, OS was censored at the date of last contact. OS was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: From first dose of study drug up to end of study (median time on study was 157.0 days, minimum of 5 days and maximum of 1320 days)
Population: The analysis population was the FAS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
days
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 123.0 [17.0 to 267.0] | 199.5 [56.0 to 905.0] | 197.5 [61.0 to 329.0] | 246.0 [190.0 to 309.0] | 214.0 [126.0 to 264.0] | 157.0 [20.0 to 218.0] | 204.0 [51.0 to 357.0]
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | NA [227.0 to NA] — Data could not be calculated due to the low number of events. | 71.5 [5.0 to 180.0] | 136.0 [14.0 to 314.0] | 144.0 [83.0 to 195.0] | 67.0 [21.0 to 336.0] | 68.0 [8.0 to 249.0] | 89.0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 149.5 [31.0 to 267.0] | 95.0 [55.0 to 195.0] | 154.0 [74.0 to 299.0] | 216.0 [161.0 to 285.0] | 176.0 [124.0 to 253.0] | 128.5 [36.0 to 199.0] | 89.0 [51.0 to 357.0]

34. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the time from the date of first dose of study drug until the date of documented relapse, treatment failure or death from any cause, whichever occurred first. For a participant with none of these events, EFS was censored at the date of last relapse-free disease assessment. A participant without post-treatment disease assessment was censored at randomization date. Treatment failure included those participants who discontinued the treatment due to "progressive disease" or "lack of efficacy" without a previous response of CR, CRp, CRi or PR. Treatment failure date referred to the start of new anti-leukemia therapy or the last treatment evaluation date when new anti-leukemia therapy date was not available. For participants who were censored, last relapse-free disease assessment date referred to the participant's last disease assessment date. EFS was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: as for outcome 33
Population: The analysis population was the FAS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 16 | 16 | 24 | 70 | 100 | 20 | 3
days
  FLT3 Mutation Positive: number analyzed (Participants) | 14 | 8 | 12 | 56 | 89 | 10 | 2
  FLT3 Mutation Positive | 52.0 [14.0 to 88.0] | 109.0 [29.0 to 357.0] | 93.5 [61.0 to 127.0] | 112.0 [92.0 to 143.0] | 121.0 [92.0 to 155.0] | 85.0 [11.0 to 157.0] | 86.0 [51.0 to 121.0]
  FLT3 Mutation Negative: number analyzed (Participants) | 2 | 8 | 12 | 14 | 11 | 10 | 1
  FLT3 Mutation Negative | 58.0 [NA to NA] — Data could not be calculated due to the low number of events. | 39.0 [5.0 to 67.0] | 74.0 [12.0 to 131.0] | 85.5 [37.0 to 126.0] | 45.0 [21.0 to 113.0] | 43.0 [8.0 to 83.0] | 71.0 [NA to NA] — Data could not be calculated due to the low number of events.
  All Participants | 58.0 [19.0 to 88.0] | 55.5 [38.0 to 92.0] | 76.0 [61.0 to 119.0] | 108.0 [90.0 to 126.0] | 118.0 [88.0 to 140.0] | 65.0 [20.0 to 100.0] | 71.0 [51.0 to 121.0]

35. Secondary Outcome: Leukemia Free Survival (LFS)
Description: LFS was defined as the time from the date of first CRc until the date of documented relapse or death for participants who achieved CRc. For a participant who was not known to have relapsed or died, LFS was censored on the date of last relapse-free disease assessment date. LFS was calculated using Kaplan-Meier method and therefore data are estimated.
Time Frame: as for outcome 33
Population: The analysis population was the FAS. Only participants who achieved CRc were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 2 | 0 | 7 | 27 | 37 | 3 | 0
days
  FLT3 Mutation Positive: number analyzed (Participants) | 1 | 0 | 5 | 26 | 36 | 3 | 0
  FLT3 Mutation Positive | 242.0 [NA to NA] — Data could not be calculated due to the low number of events. |  | 98.0 [56.0 to 1126.0] | 98.0 [58.0 to 187.0] | 146.0 [47.0 to 247.0] | 296.0 [130.0 to 462.0] |
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 0 | 2 | 1 | 1 | 0 | 0
  FLT3 Mutation Negative | NA [NA to NA] — Data could not be calculated due to the low number of events. |  | 41.0 [22.0 to 60.0] | 99.0 [NA to NA] — Data could not be calculated due to the low number of events. | 38.0 [NA to NA] — Data could not be calculated due to the low number of events. |  |
  All Participants | 242.0 [NA to NA] — Data could not be calculated due to the low number of events. |  | 79.0 [22.0 to 1126.0] | 98.0 [58.0 to 187.0] | 146.0 [45.0 to 247.0] | 296.0 [130.0 to 462.0] |

36. Secondary Outcome: Percentage of Participants Who Achieved Transfusion Conversion
Description: Participants who achieved transfusion conversion were defined as the number of participants who were transfusion dependent at baseline period but became transfusion independent at post-baseline period divided by the total number of participants who were transfusion dependent at baseline period. Participants were considered baseline transfusion dependent if there were RBC or platelet transfusions within the baseline period. Participants were considered post-baseline transfusion independent if they were on treatment >=84 days, and if there was one consecutive 56 days without any RBC or platelet transfusion within post-baseline period. If participants were on treatment >28 days but <84 days, and there was no RBC or platelet transfusion within post-baseline period, or on treatment <=28 days, post-baseline transfusion status was not evaluable. Exact 95% confidence interval was estimated using the binomial distribution.
Time Frame: Baseline (28 days prior to first dose until 28 days after the first dose) and postbaseline (from 29 days after first dose date until last dose date); median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days
Population: The analysis population was the FAS. Participants who were transfusion dependent at baseline and had evaluable post-baseline transfusion status were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 7 | 8 | 16 | 49 | 63 | 8 | 2
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 6 | 5 | 8 | 40 | 57 | 4 | 1
  FLT3 Mutation Positive | 0 [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | 0 [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | 37.5 [8.5 to 75.5] | 27.5 [14.6 to 43.9] | 40.4 [27.6 to 54.2] | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline.
  FLT3 Mutation Negative: number analyzed (Participants) | 1 | 3 | 8 | 9 | 6 | 4 | 1
  FLT3 Mutation Negative | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | 12.5 [0.3 to 52.7] | 22.2 [2.8 to 60.0] | 33.3 [4.3 to 77.7] | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline.
  All Participants | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | 25.0 [7.3 to 52.4] | 26.5 [14.9 to 41.1] | 39.7 [27.6 to 52.8] | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline. | NA [NA to NA] — No data could be calculated due to the low number of participants who had evaluable transfusion status postbaseline.

37. Secondary Outcome: Percentage of Participants Who Achieved Transfusion Maintenance
Description: Participants who achieved transfusion maintenance were defined as the number of participants who were transfusion independent at baseline period and still maintained transfusion independent at post-baseline period divided by the total number of participants who were transfusion independent at baseline period.
Time Frame: as for outcome 36
Population: The analysis population was the FAS. Participants who were transfusion independent at baseline and had evaluable post-baseline transfusion status were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 20 mg | Gilteritinib 40 mg | Gilteritinib 80 mg | Gilteritinib 120 mg | Gilteritinib 200 mg | Gilteritinib 300 mg | Gilteritinib 450 mg
Number analyzed (Participants) | 0 | 0 | 1 | 7 | 10 | 0 | 1
percentage of participants
  FLT3 Mutation Positive: number analyzed (Participants) | 0 | 0 | 1 | 4 | 10 | 0 | 1
  FLT3 Mutation Positive |  |  | 100.0 [2.5 to 100] | 75.0 [19.4 to 99.4] | 80.0 [44.4 to 97.5] |  | 100.0 [2.5 to 100.0]
  FLT3 Mutation Negative: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 0 | 0
  FLT3 Mutation Negative |  |  |  | 33.3 [0.8 to 90.6] |  |  |
  All Participants |  |  | 100.0 [2.5 to 100.0] | 57.1 [18.4 to 90.1] | 80.0 [44.4 to 97.5] |  | 100.0 [2.5 to 100.0]

38. Secondary Outcome: AUC24 of Gilteritinib in Co-administration With Voriconazole
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (gilteritinib)
Population: The analysis population was the PKAS, with participants administered 20 mg gilteritinib and voriconazole.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 20 mg in Expansion Phase
Number analyzed (Participants) | 1
ng*h/mL | 919.3 (NA) — SD could not be calculated due to a sample size of 1.

39. Secondary Outcome: Cmax of Gilteritinib in Co-administration With Voriconazole
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (gilteritinib)
Population: The analysis population was the PKAS, with participants administered 20 mg gilteritinib and voriconazole.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 20 mg in Expansion Phase
Number analyzed (Participants) | 1
ng/mL | 63.79 (NA) — SD could not be calculated due to a sample size of 1.

40. Secondary Outcome: AUClast of Gilteritinib in Co-administration With Voriconazole
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (gilteritinib)
Population: The analysis population was the PKAS, with participants administered 20 mg gilteritinib and voriconazole.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 20 mg in Expansion Phase
Number analyzed (Participants) | 1
ng*h/mL | 919.3 (NA) — SD could not be calculated due to a sample size of 1.

41. Secondary Outcome: Tmax of Gilteritinib in Co-administration With Voriconazole
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (gilteritinib)
Population: The analysis population was the PKAS, with participants administered 20 mg gilteritinib and voriconazole.
Measure: Median (Full Range); unit: hours
Arm/Group | Gilteritinib 20 mg in Expansion Phase
Number analyzed (Participants) | 1
hours | 2.08 [2.08 to 2.08]

42. Secondary Outcome: AUC24 of Midazolam Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
ng*h/mL
  Midazolam Alone (Day -1): number analyzed (Participants) | 15
  Midazolam Alone (Day -1) | 66.55 (57.70)
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 8
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 81.56 (65.84)
Statistical Analysis 1: Comparison: Gilteritinib 300 mg in Expansion Phase; Statistical Comparison of Midazolam Exposure after Administration of Midazolam Alone or Coadministered with Gilteritinib: The difference of least squares (LS) means of log-transformed pharmacokinetic parameters between midazolam alone and midazolam + gilteritinib and its 90% CI are backtransformed to the raw scale and are expressed as percent; Test type: Other; Geometric LS Mean Ratio = 109.46, 90% CI 2-sided [49.82 to 240.48]

43. Secondary Outcome: AUC24 of Metabolite 1-Hydroxymidazolam After Administration of Midazolam With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
ng*h/mL
  Midazolam Alone (Day -1): number analyzed (Participants) | 15
  Midazolam Alone (Day -1) | 20.44 (24.80)
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 8
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 23.10 (21.64)
Statistical Analysis 1: Comparison: Gilteritinib 300 mg in Expansion Phase; Statistical Comparison of Midazolam Exposure after Administration of Midazolam Alone or Coadministered with Gilteritinib: The difference of LS means of log-transformed pharmacokinetic parameters between 1-hydroxymidazolam alone and 1-hydroxymidazolam + gilteritinib and its 90% CI are backtransformed to the raw scale and are expressed as percent; Test type: Other; Geometric LS Mean Ratio = 149.90, 90% CI [74.88 to 300.06]

44. Secondary Outcome: Cmax of Midazolam Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
ng/mL
  Midazolam Alone (Day -1): number analyzed (Participants) | 16
  Midazolam Alone (Day -1) | 14.68 (8.923)
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 9
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 18.45 (9.452)
Statistical Analysis 1: Comparison: Gilteritinib 300 mg in Expansion Phase; Statistical Comparison of Midazolam Exposure after Administration of Midazolam Alone or Coadministered with Gilteritinib: The difference of LS means of log-transformed pharmacokinetic parameters between midazolam alone and midazolam + gilteritinib and its 90% CI are backtransformed to the raw scale and are expressed as percent; Test type: Other; Geometric LS Mean Ratio = 111.64, 90% CI 2-sided [69.54 to 179.25]

45. Secondary Outcome: Cmax of 1-Hydroxymidazolam After Administration of Midazolam With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
ng/mL
  Midazolam Alone (Day -1): number analyzed (Participants) | 16
  Midazolam Alone (Day -1) | 4.562 (2.858)
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 9
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 5.053 (3.158)
Statistical Analysis 1: Comparison: Gilteritinib 300 mg in Expansion Phase; Statistical Comparison of Midazolam Exposure after Administration of Midazolam Alone or Coadministered with Gilteritinib: The difference of LS means of log-transformed pharmacokinetic parameters between 1-hydroxymidazolam/midazolam alone and 1-hydroxymidazolam/midazolam + gilteritinib and its 90% CI are backtransformed to the raw scale and are expressed as percent; Test type: Other; Geometric LS Mean Ratio = 123.47, 90% CI 2-sided [72.41 to 210.52]

46. Secondary Outcome: AUClast of Midazolam Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
ng*h/mL
  Midazolam Alone (Day -1): number analyzed (Participants) | 16
  Midazolam Alone (Day -1) | 59.48 (59.49)
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 9
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 82.44 (64.25)

47. Secondary Outcome: AUClast of 1-Hydroxymidazolam After Administration of Midazolam With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
ng*h/mL
  Midazolam Alone (Day -1): number analyzed (Participants) | 16
  Midazolam Alone (Day -1) | 17.05 (24.70)
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 9
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 23.58 (22.07)

48. Secondary Outcome: Tmax of Midazolam Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Median (Full Range); unit: hours
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
hours
  Midazolam Alone (Day -1): number analyzed (Participants) | 16
  Midazolam Alone (Day -1) | 0.5000 [0.367 to 2.00]
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 9
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 1.00 [0.317 to 4.13]

49. Secondary Outcome: Tmax of 1-Hydroxymidazolam After Administration of Midazolam With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 2, 4, 6, 24 hours postdose (midazolam)
Population: The analysis population was the PKAS, with participants administered 300 mg gilteritinib and midazolam.
Measure: Median (Full Range); unit: hours
Arm/Group | Gilteritinib 300 mg in Expansion Phase
Number analyzed (Participants) | 17
hours
  Midazolam Alone (Day -1): number analyzed (Participants) | 16
  Midazolam Alone (Day -1) | 0.5583 [0.483 to 2.00]
  Midazolam + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 9
  Midazolam + Gilteritinib (Cycle 1 Day 15) | 1.00 [0.317 to 4.13]

50. Secondary Outcome: Area Under the Concentration-time Curve From the Time of Dosing Extrapolated to Time Infinity (AUCinf) of Cephalexin Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
ng*h/mL
  Cephalexin Alone (Day -1): number analyzed (Participants) | 18
  Cephalexin Alone (Day -1) | 57650 (20386)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 13
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 51873 (18819)
Statistical Analysis 1: Comparison: Gilteritinib 200 mg in Expansion Phase; Statistical Assessment of the Effect of Gilteritinib on Cephalexin Pharmacokinetics after Administration of Cephalexin Alone or Coadministered with Gilteritinib: The difference of LS means of log-transformed pharmacokinetic parameters between cephalexin alone and cephalexin + gilteritinib and its 90% CI are backtransformed to the raw scale and are expressed as percent; Test type: Other; Geometric LS Mean Ratio = 93.96, 90% CI 2-sided [75.29 to 117.26]

51. Secondary Outcome: Cmax of Cephalexin Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
ng/mL
  Cephalexin Alone (Day -1): number analyzed (Participants) | 20
  Cephalexin Alone (Day -1) | 17688 (6680)
  Cephalexin + Gilteritinib (Cycle 1 day 15): number analyzed (Participants) | 16
  Cephalexin + Gilteritinib (Cycle 1 day 15) | 16075 (4606)
Statistical Analysis 1: Comparison: Gilteritinib 200 mg in Expansion Phase; [analysis description as in outcome 50, analysis 1]; Test type: Other; Geometric LS Mean Ratio = 91.46, 90% CI 2-sided [74.60 to 112.12]

52. Secondary Outcome: AUClast of Cephalexin Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
ng*h/mL
  Cephalexin Alone (Day -1): number analyzed (Participants) | 20
  Cephalexin Alone (Day -1) | 53183 (26877)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 16
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 54963 (29531)
Statistical Analysis 1: Comparison: Gilteritinib 200 mg in Expansion Phase; [analysis description as in outcome 50, analysis 1]; Test type: Other; Geometric LS Mean Ratio = 97.71, 90% CI 2-sided [74.19 to 128.70]

53. Secondary Outcome: Tmax of Cephalexin Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Median (Full Range); unit: hours
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
hours
  Cephalexin Alone (Day -1): number analyzed (Participants) | 20
  Cephalexin Alone (Day -1) | 1.500 [1.00 to 4.02]
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 16
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 1.483 [1.00 to 5.88]

54. Secondary Outcome: T1/2 of Cephalexin Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
hours
  Cephalexin Alone (Day -1): number analyzed (Participants) | 18
  Cephalexin Alone (Day -1) | 1.822 (0.5914)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 13
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 1.827 (0.7175)

55. Secondary Outcome: Apparent Total Systemic Clearance After Single or Multiple Extravascular Dosing (CL/F) of Cephalexin Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
L/h
  Cephalexin Alone (Day -1): number analyzed (Participants) | 18
  Cephalexin Alone (Day -1) | 9.713 (3.319)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 13
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 10.58 (2.977)
Statistical Analysis 1: Comparison: Gilteritinib 200 mg in Expansion Phase; [analysis description as in outcome 50, analysis 1]; Test type: Other; Geometric LS Mean Ratio = 106.42, 90% CI 2-sided [85.28 to 132.81]

56. Secondary Outcome: Apparent Volume of Distribution During the Terminal Elimination Phase After Single Extravascular Dosing (Vz/F) of Cephalexin Administered With and Without Gilteritinib
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
liters
  Cephalexin Alone (Day -1): number analyzed (Participants) | 18
  Cephalexin Alone (Day -1) | 24.07 (7.173)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 13
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 25.86 (5.346)

57. Secondary Outcome: Amount of Drug Excreted in Urine (Aelast) of Cephalexin Administered With and Without Gilteritinib
Description: Urine samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: 0-3 hours, 3-6 hours, 6-24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
mg
  Cephalexin Alone (Day -1): number analyzed (Participants) | 13
  Cephalexin Alone (Day -1) | 548.9 (523.7)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 10
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 448.8 (306.1)
Statistical Analysis 1: Comparison: Gilteritinib 200 mg in Expansion Phase; [analysis description as in outcome 50, analysis 1]; Test type: Other; Geometric LS Mean Ratio = 83.93, 90% CI 2-sided [46.53 to 151.39]

58. Secondary Outcome: Fraction of Drug Excreted Into Urine in Percentage (%Ae) of Cephalexin Administered With and Without Gilteritinib
Description: Urine samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: 0-3 hours, 3-6 hours, 6-24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
percentage
  Cephalexin Alone (Day -1): number analyzed (Participants) | 13
  Cephalexin Alone (Day -1) | 109.8 (104.7)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 10
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 89.75 (61.21)

59. Secondary Outcome: Renal Clearance (CLr) of Cephalexin in Administered With and Without Gilteritinib
Description: Urine samples were used for pharmacokinetic assessments.
Time Frame: Day -1 and cycle 1 day 15: 0-3 hours, 3-6 hours, 6-24 hours postdose (cephalexin)
Population: The analysis population was the PKAS, with participants administered 200 mg gilteritinib and cephalexin.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Gilteritinib 200 mg in Expansion Phase
Number analyzed (Participants) | 100
L/h
  Cephalexin Alone (Day -1): number analyzed (Participants) | 13
  Cephalexin Alone (Day -1) | 8.784 (8.727)
  Cephalexin + Gilteritinib (Cycle 1 Day 15): number analyzed (Participants) | 6
  Cephalexin + Gilteritinib (Cycle 1 Day 15) | 11.04 (8.430)
Statistical Analysis 1: Comparison: Gilteritinib 200 mg in Expansion Phase; [analysis description as in outcome 50, analysis 1]; Test type: Other; Geometric LS Mean Ratio = 82.84, 90% CI 2-sided [40.25 to 170.48]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (median treatment duration was 69.5 days, minimum of 3 days and maximum of 1320 days)
Description: The total number of deaths (all causes) includes deaths reported after the time frame above.
Groups:
- Gilterinib 20 mg in Escalation Phase: Participants received a single dose of 20 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 20 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
- Gilterinib 40 mg in Escalation Phase: Participants received a single dose of 40 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 40 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
- Gilterinib 80 mg in Escalation Phase: Participants received a single dose of 80 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 80 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
- Gilterinib 120 mg in Escalation Phase: Participants received a single dose of 120 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 120 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
- Gilterinib 200 mg in Escalation Phase: Participants received a single dose of 200 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 200 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
- Gilterinib 300 mg in Escalation Phase: Participants received a single dose of 300 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 300 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
- Gilterinib 450 mg in Escalation Phase: Participants received a single dose of 450 mg gilteritinib orally on day -2 to evaluate pharmacokinetics of gilteritinib. Then starting on day 1 of cycle 1, participants received 450 mg gilteritinib orally once daily in 28-day cycles until disease progression or participant discontinuation in the escalation phase of the study.
- Gilterinib 20 mg in Expansion Phase: Participants received 20 mg gilteritinib orally once daily stating on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. Starting on day 16 of cycle 1, participants also received 200 mg voriconazole orally every 12 hours through day 1 of cycle 2.
- Gilterinib 40 mg in Expansion Phase: Participants received 40 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
- Gilterinib 80 mg in Expansion Phase: Participants received 80 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
- Gilterinib 120 mg in Expansion Phase: Participants received 120 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study.
- Gilterinib 200 mg in Expansion Phase: Participants received 200 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. On day -1 and day 15 of cycle 1, certain participants also received 500 mg cephalexin as a single oral dose.
- Gilterinib 300 mg in Expansion Phase: Participants received 300 mg gilteritinib orally once daily starting on day 1 of cycle 1 and continued in 28-day cycles until disease progression or participant discontinuation in the expansion phase of the study. On day -1 and day 15 of cycle 1, participants also received 2 mg midazolam as a single oral dose.
Arm/Group | Gilterinib 20 mg in Escalation Phase | Gilterinib 40 mg in Escalation Phase | Gilterinib 80 mg in Escalation Phase | Gilterinib 120 mg in Escalation Phase | Gilterinib 200 mg in Escalation Phase | Gilterinib 300 mg in Escalation Phase | Gilterinib 450 mg in Escalation Phase | Gilterinib 20 mg in Expansion Phase | Gilterinib 40 mg in Expansion Phase | Gilterinib 80 mg in Expansion Phase | Gilterinib 120 mg in Expansion Phase | Gilterinib 200 mg in Expansion Phase | Gilterinib 300 mg in Expansion Phase
All-Cause Mortality (participants affected / at risk) | 4/5 | 2/3 | 3/3 | 3/3 | 2/3 | 3/3 | 3/3 | 10/12 | 13/13 | 21/21 | 53/66 | 82/100 | 16/17
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/3 | 2/3 | 1/3 | 2/3 | 2/3 | 2/3 | 8/12 | 12/13 | 19/21 | 52/66 | 92/100 | 14/17
Other Adverse Events (participants affected / at risk) | 5/5 | 2/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 12/12 | 12/13 | 20/21 | 62/66 | 97/100 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilterinib 20 mg in Escalation Phase (N=5) | Gilterinib 40 mg in Escalation Phase (N=3) | Gilterinib 80 mg in Escalation Phase (N=3) | Gilterinib 120 mg in Escalation Phase (N=3) | Gilterinib 200 mg in Escalation Phase (N=3) | Gilterinib 300 mg in Escalation Phase (N=3) | Gilterinib 450 mg in Escalation Phase (N=3) | Gilterinib 20 mg in Expansion Phase (N=12) | Gilterinib 40 mg in Expansion Phase (N=13) | Gilterinib 80 mg in Expansion Phase (N=21) | Gilterinib 120 mg in Expansion Phase (N=66) | Gilterinib 200 mg in Expansion Phase (N=100) | Gilterinib 300 mg in Expansion Phase (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (6) | 2 (5) | 0 (0) | 4 (6) | 7 (7) | 5 (11) | 18 (28) | 35 (58) | 4 (4)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 5 (5) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (4) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 4 (6) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 9 (13) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute graft versus host disease in intestine (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 2 (2) | 5 (7) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (10) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 13 (15) | 12 (15) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 10 (10) | 19 (25) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 4 (6) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinusitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (4) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 5 (8) | 9 (10) | 20 (25) | 4 (5)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (4) | 5 (5) | 14 (16) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute promyelocytic leukaemia differentiation syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 11 (13) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis deep (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilterinib 20 mg in Escalation Phase (N=5) | Gilterinib 40 mg in Escalation Phase (N=3) | Gilterinib 80 mg in Escalation Phase (N=3) | Gilterinib 120 mg in Escalation Phase (N=3) | Gilterinib 200 mg in Escalation Phase (N=3) | Gilterinib 300 mg in Escalation Phase (N=3) | Gilterinib 450 mg in Escalation Phase (N=3) | Gilterinib 20 mg in Expansion Phase (N=12) | Gilterinib 40 mg in Expansion Phase (N=13) | Gilterinib 80 mg in Expansion Phase (N=21) | Gilterinib 120 mg in Expansion Phase (N=66) | Gilterinib 200 mg in Expansion Phase (N=100) | Gilterinib 300 mg in Expansion Phase (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 4 (4) | 7 (10) | 27 (84) | 33 (65) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 7 (8) | 15 (20) | 3 (3)
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 4 (6) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (28) | 12 (29) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 12 (27) | 19 (44) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 6 (7) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 12 (13) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (10) | 6 (7) | 0 (0)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (9) | 0 (0)
Retinal exudates (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (8) | 6 (6) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 15 (19) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 5 (5) | 12 (14) | 32 (36) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 2 (2) | 5 (12) | 27 (44) | 45 (71) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 10 (10) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 6 (8) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 8 (9) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 4 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (5) | 15 (22) | 28 (37) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (3) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 8 (9) | 14 (15) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 5 (6) | 13 (16) | 22 (31) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 6 (8) | 19 (20) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 12 (15) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (6) | 1 (2) | 1 (3) | 4 (5) | 5 (6) | 8 (11) | 27 (38) | 32 (47) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 5 (5) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (5) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 11 (13) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 3 (5) | 6 (7) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 5 (11) | 17 (22) | 31 (48) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 6 (9) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (4) | 4 (6) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 18 (25) | 24 (33) | 3 (3)
Serositis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 6 (12) | 0 (0)
Graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (6) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Laryngitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (6) | 5 (6) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 7 (9) | 5 (11) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 5 (7) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 3 (4) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 10 (11) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 11 (15) | 18 (22) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 3 (9) | 16 (26) | 25 (46) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (3) | 1 (1) | 3 (9) | 20 (33) | 35 (61) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (12) | 10 (12) | 15 (19) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 3 (3) | 1 (1) | 12 (22) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 15 (27) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (9) | 13 (23) | 19 (40) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 7 (9) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chest X-ray abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (13) | 9 (11) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 4 (7) | 5 (7) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 8 (16) | 14 (29) | 0 (0)
Platelet count decreased (Investigations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (8) | 3 (4) | 1 (1) | 12 (26) | 17 (37) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 5 (6) | 1 (1)
Ultrasound liver abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volume blood increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 6 (7) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 12 (18) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (14) | 13 (30) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 11 (13) | 19 (21) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 10 (10) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 14 (16) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 5 (6) | 9 (10) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 10 (11) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 4 (15) | 7 (15) | 18 (28) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (17) | 11 (23) | 23 (50) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (9) | 2 (3) | 2 (11) | 10 (20) | 25 (33) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 13 (19) | 17 (25) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (8) | 8 (16) | 20 (26) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (10) | 11 (13) | 2 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 12 (15) | 16 (23) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 8 (9) | 9 (11) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 4 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 12 (14) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 10 (13) | 11 (15) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 17 (19) | 26 (34) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 9 (10) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 9 (9) | 11 (12) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 10 (14) | 14 (20) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 7 (9) | 5 (6) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 7 (12) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (8) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 6 (6) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (7) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 6 (6) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 4 (4) | 10 (12) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (6) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 8 (9) | 13 (14) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 7 (8) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 6 (6) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 4 (5) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 7 (8) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 7 (7) | 18 (27) | 26 (29) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (5) | 4 (5) | 19 (23) | 28 (38) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 16 (18) | 20 (24) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (8) | 11 (14) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 9 (9) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 5 (6) | 8 (11) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 10 (14) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 3 (3) | 3 (5) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 8 (8) | 1 (1)
Eccrine squamous syringometaplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 4 (4) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 4 (4) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 7 (12) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 11 (11) | 11 (13) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 7 (9) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 2 (4)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (8) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 7 (7) | 16 (34) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 10 (11) | 25 (32) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 8 (8) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT02014558/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT02014558/SAP_001.pdf